CLINICAL TRIAL: NCT03980444
Title: Determine the Effectiveness of Convective Uses of Basket Wires for the Maintenance of Stone and Pneumatic Probe in the Treatment of Ureteral Stones
Brief Title: Effectiveness Basket Wires for the Maintenance of Stone and Pneumatic Probe in the Treatment of Ureteral Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Sadegh Bagheri Baghdasht (Other)
Responsible Party: Sponsor-Investigator, Mohammad Sadegh Bagheri Baghdasht, student research committee, Baqiyatallah Medical Sciences University
Organization: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.BMSU.REC.1393.4
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Ureter Stone
Keywords: Ureterolithiasis; Manganese Poisoning; Lithotripsy; Ureteroscopy; stone baske
MeSH Terms: conditions — Ureterolithiasis; Manganese Poisoning | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients included in the study included the necessary tests U/A, K, Na, Cr, BUN, CBC, And U / C was checked and anesthesia counseling was done. The demographic and clinical data of the patients were recorded.
  Then patients as random allocation were divided into two groups: A (control group) and group B (use of a pneumatic basket of wire). The dividing person and the patients themselves were not aware of which group they were in.
  In each group, ureteroscopy was performed using a standard F9.5 ureteroscope. After reaching the rock in group A, the probe of the pneumatic crusher was passed through the working channel of the ureteroscope and began crushing the rock.
  In group B (using a basket of wires3F) the helical type was passed through the four wires of the working channel of the orthoscope and routed to the proximal part of the rock, and the stone was routed to the bowl, then the stone was ducted The gasket was kept, and the same as A group.
Who Masked: Investigator
Masking Description: patients as random allocation were divided into two groups: A (control group, no basket of bases and group B (use of pneumatic synchronous buccal waist). The dividing person and the patients themselves were not aware of which group they were in. They were double-blind Was.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group, no basket of wire (Experimental): The dividing person and the patients themselves were not aware of which group they were in. They were double-blind Was.
  In each group, ureteroscopy was performed using a standard F9.5 ureteroscope. After reaching the rock in group A (control), the probe of the pneumatic crusher was passed through the working channel of the ureteroscope and began crushing the rock.
  During the crushing process, the minimum flow of water, flattening and the single-shot impact was used to minimize the stone's retropulsion.
  Interventions: Procedure: control group, no basket
- using a basket of wires (Sham Comparator): In group B (using a basket of wires3F) the helical type was passed through the four wires of the working channel of the orthoscope and routed to the proximal part of the rock, and the stone was routed to the bowl, then the stone was ducted The gasket was kept, and the probe of the pneumatic crusher also passed through the working channel and proceeded to break it down. Conditions were observed during the stomach as control group. Urethroscopic crushing was performed by a urologist in both groups under similar technical conditions. Findings during and after the completion of crushing include the success, stone retropulsion or parts larger than 3 mm, which requires secondary measures (SWL - ureter stenting, resection ureteroscopy), the duration of stone breakdown and traumatic ureteric complications in both groups it is registered
  Interventions: Device: Basket of wire

INTERVENTIONS:
Device: Basket of wire — (using a basket of wires3F) the helical type was passed through the four wires of the working channel of the orthoscope and routed to the proximal part of the rock, and the stone was routed to the bowl, then the stone was ducted The gasket was kept, and the probe of the pneumatic crusher also passed through the working channel and proceeded to break it down. Conditions were observed during the stomach as control group. Urethroscopic crushing was performed by a urologist in both groups under similar technical conditions. Findings during and after the completion of crushing include the success, stone retropulsion or parts larger than 3 mm, which requires secondary measures (SWL - ureter stenting, resection ureteroscopy), the duration of stone breakdown and traumatic ureteric complications in both groups it is registered
  Arms: using a basket of wires
Procedure: control group, no basket — In each group, ureteroscopy was performed using a standard F9.5 ureteroscope. After reaching the rock in group A (control), the probe of the pneumatic crusher was passed through the working channel of the ureteroscope and began crushing the rock.
  During the crushing process, the minimum flow of water, flattening and the single-shot impact was used to minimize the stone's retropulsion.
  Arms: control group, no basket of wire

SUMMARY:
Patients included in the study included the necessary tests U / A, K, Na, Cr, BUN, CBC, And U / C was checked and anesthesia counseling was done. Patients were prepared for action. The demographic and clinical data of the patients, including age, sex, size, and location of the stones were recorded.

Then patients as random allocation were divided into two groups: A (control group, no basket of bases and group B (use of pneumatic synchronous buccal waist). The dividing person and the patients themselves were not aware of which group they were in. They were double-blind was.

In each group, ureteroscopy was performed using a standard F9.5 ureteroscope. After reaching the rock in group A (control), the probe of the pneumatic crusher was passed through the working channel of the ureteroscope and began crushing the rock.

During the crushing process, the minimum flow of water, flattening and the single-shot impact was used to minimize the stone's retropulsion.

In group B (using a basket of wires3F) the helical type was passed through the four wires of the working channel of the ureteroscope and routed to the proximal part of the rock, and the stone was routed to the bowl, then the stone was ducted The gasket was kept, and the probe of the pneumatic crusher also passed through the working channel and proceeded to break it down. Conditions were observed during the stomach as the control group. Ureteroscopic crushing was performed by a urologist in both groups under similar technical conditions. Findings during and after the completion of crushing include the success, stone retropulsion or parts larger than 3 mm, which requires secondary measures (SWL - ureter stenting, resection ureteroscopy), the duration of stone breakdown and traumatic ureteric complications in both groups it is registered.

ELIGIBILITY:
Inclusion Criteria:

* Individual interest in engaging in research
* Patients with ureter stones
* Symptoms of severe and resistant to supportive and therapeutic treatment
* Ureteral stones cause ureteral obstruction
* Ureteral stones, which is not likely to be disposed of by duration and size, have been selected for ureteroscopic lithotripsy.

Exclusion Criteria:

* Patients with urinary tract infection
* Not having a proper cardiovascular condition and not approved by a cardiologist or anesthetist
* Patients who are dissatisfied with ureteroscopic crushing and patients who do not have access to rocks during ureteroscopic surgery
* Individual interest in leaving the study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Stone size | 24 hours
  The largest diameter of the stone in the imaging of millimeters
Crushing time | up to 23minute
  Duration needed to break the stone to the minute
Demographic questionnaire | 24 hours
  The demographic questionnaire was used to collect information
Troma in the ureter area | up to 24 hours
  Follow up of patients for perforation, missing stone, and ureter ligation according to observations during and after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - MS Bagheri-baghdasht, Tehran
  - MS bagheri-baghdast, Tehran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elashry OM, Tawfik AM. Preventing stone retropulsion during intracorporeal lithotripsy. Nat Rev Urol. 2012 Dec;9(12):691-8. doi: 10.1038/nrurol.2012.204. Epub 2012 Nov 20. PMID 23165399
- [Result] Rane A, Bradoo A, Rao P, Shivde S, Elhilali M, Anidjar M, Pace K, D'A Honey JR. The use of a novel reverse thermosensitive polymer to prevent ureteral stone retropulsion during intracorporeal lithotripsy: a randomized, controlled trial. J Urol. 2010 Apr;183(4):1417-21. doi: 10.1016/j.juro.2009.12.023. Epub 2010 Feb 20. PMID 20171695
- [Result] Vejdani K, Eisner BH, Pengune W, Stoller ML. Effect of laser insult on devices used to prevent stone retropulsion during ureteroscopic lithotripsy. J Endourol. 2009 Feb;23(2):249-51. doi: 10.1089/end.2008.0352. PMID 19220084
- [Result] Ursiny M, Eisner BH. Cost-effectiveness of anti-retropulsion devices for ureteroscopic lithotripsy. J Urol. 2013 May;189(5):1762-6. doi: 10.1016/j.juro.2012.11.085. Epub 2012 Nov 15. PMID 23159589
- [Result] Wu JA, Ngo TC, Hagedorn JC, Macleod LC, Chung BI, Shinghal R. The accordion antiretropulsive device improves stone-free rates during ureteroscopic laser lithotripsy. J Endourol. 2013 Apr;27(4):438-41. doi: 10.1089/end.2012.0332. Epub 2013 Feb 6. PMID 23387558
- [Result] Pagnani CJ, El Akkad M, Bagley DH. Prevention of stone migration with the Accordion during endoscopic ureteral lithotripsy. J Endourol. 2012 May;26(5):484-8. doi: 10.1089/end.2011.0386. Epub 2012 Jan 4. PMID 22192096
- [Result] Farahat YA, Elbahnasy AE, Elashry OM. A randomized prospective controlled study for assessment of different ureteral occlusion devices in prevention of stone migration during pneumatic lithotripsy. Urology. 2011 Jan;77(1):30-5. doi: 10.1016/j.urology.2010.05.063. Epub 2010 Oct 20. PMID 20970173